CLINICAL TRIAL: NCT04209569
Title: One Nutrition in Complex Environments (ONCE), a Cluster-randomized Trial of Nutrition Education and Access to Simple Supportive Technologies in Improving Agricultural Practices and Water Quality Management
Brief Title: One Nutrition in Complex Environments (ONCE)
Acronym: ONCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: GOAL, Ireland (Unknown); Centro Internacional de Mejoramiento de Maiz y Trigo Internacional, Mexico (Unknown); Cornell University (Other)
Responsible Party: Principal Investigator, Shibani Ghosh, Research Associate Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13426
Record Dates: First submitted 2019-12-08; First posted 2019-12-24 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Nutrition Poor; Aflatoxins Toxicity; Water-Related Diseases
Keywords: SBCC; child wasting; aflatoxin; coliform; Uganda
MeSH Terms: conditions — Malnutrition; Waterborne Diseases

STUDY DESIGN:
Intervention Model Description: The study design is a three-arm cluster randomized controlled superiority design (cRCT) with a 1:1:1 allocation ratio. The study arms will be: Group 1: NIPP arm; Group 2: NIPP+ arm; and Group 3: Non-intervention control arm.
  for the venous aflatoxin sub-study, 36 women will be purposively selected from the eligible communities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NIPP (Active Comparator): The NIPP group is a standard social behavior change (SBCC) intervention that tackles a set of underlying causes of malnutrition, with the potential to have both a curative and preventative impact on child malnutrition. The approach in this group/arm involves training and pragmatic behavior change education reinforced by practical activities over a 12-week period to both men and women in selected communities. It aims to utilize easy, viable and accessible solutions within the community that can be used to improve and protect household health and nutrition. The 12-week lesson plans for the circles are divided into 3 components, i) hands-on behavior change sessions that focus on the key pre-identified causes of malnutrition to improve awareness and practice ii) micro-gardening for improved household nutrition security and iii) participatory cooking demonstrations to stimulate improvements in nutritional status and care practices.
  Interventions: Behavioral: Nutrition Impact and Positive Practice Circle (NIPP)
- NIPP+ (Experimental): In addition to establishing the circles and implementing the three NIPP components also implemented in the NIPP arm, those randomized to the NIPP+ arm will be provided access to innovations to allow and encourage the households and communities to translate the knowledge into positive practices. The innovations and access to vendors who sell innovations will be made available during the training to the NIPP+ volunteers who will provide trainings and access to vendors during the circle meetings. Most of the additions will be made accessible at a subsidized/low cost. The NIPP+ officers from the program will support NIPP+ volunteers in collaboration with agricultural extension officers.
  Interventions: Behavioral: Nutrition Impact and Positive Practice Circle (NIPP)
- Control (No Intervention): No Intervention

INTERVENTIONS:
Behavioral: Nutrition Impact and Positive Practice Circle (NIPP) — GOAL's NIPP approach is a gendered, grass-roots SBC approach, tackling a package of underlying behavioral determinants of malnutrition, irrespective of the particular manifestation. The approach is multi-sectoral in nature. It also has a strong monitoring, evaluation and adaptive learning component by design. The intervention approach (based on GOAL's NIPP approach) involves the creation of community, male and female circles in each community with messaging and activities targeted towards the three groups in varying intensities. While the male and female circles meet 2-3 times per week for a maximum period of 12 weeks while the community circles will meet for approximately three hours at any one time over a period of 2-7 days. (See GOAL NIPP Implementation Guidelines)
  Arms: NIPP; NIPP+

SUMMARY:
This study asks the research question "Does enabling families (particularly mothers and other caregivers) to 'assess and act' on drivers of malnutrition through a targeted SBC+ package succeed in a sustained reduction of risk factors thereby improving child health and nutrition?" This study aims to implement and measure the effects of a multi-level multi-sectoral behavior change information intervention in Agago District of Northern Uganda and determine potential for scale up in a complex environment.

The study design is a three-arm cluster randomized controlled superiority design (cRCT) with a 1:1:1 allocation ratio. The study arms will be: Group 1: NIPP arm; Group 2: NIPP+ arm; and Group 3: Non-intervention control arm. A barrier analysis will be conducted to ensure appropriate targeting and contextualization of the NIPP and NIPP+ approaches prior to implementation. Each intervention arm will receive a 12-week intervention (NIPP or NIPP+) with active monitoring and longitudinal follow ups post intervention at 2, 6, and 12-months post-intervention. The total sample size for the Barrier Analysis will be a maximum of 450 caregivers; for the main intervention, 900 households (300/arm) will be purposely sampled from the randomly selected communities. Respondents for the qualitative portion will be purposely selected.

DETAILED DESCRIPTION:
Objective: This study asks the research question "Does enabling families (particularly mothers and other caregivers) to 'assess and act' on drivers of malnutrition through a targeted SBC+ package succeed in a sustained reduction of risk factors thereby improving child health and nutrition?" This study aims to implement and measure the effects of a multi-level multi-sectoral behavior change information intervention in Agago District of Northern Uganda and determine potential for scale up in a complex environment.

Intervention: Through a collaboration between Tufts University, GOAL International, CIMMYT, and Cornell University, GOAL will implement Nutrition Impact and Positive Practice (NIPP) circles as the standard SBC intervention against which the hypotheses will be tested. GOAL will also implement a NIPP+ approach which will integrate additional interventions for water, sanitation, and hygiene (WASH), and use of improved agriculture inputs. These interventions will be measured by outcome indicators measuring aflatoxin exposure, water contamination, and knowledge transferred to action.

Design: The study design is a three-arm cluster randomized controlled superiority design (cRCT) with a 1:1:1 allocation ratio. The study arms will be: Group 1: NIPP arm; Group 2: NIPP+ arm; and Group 3: Non-intervention control arm. A barrier analysis will be conducted to ensure appropriate targeting and contextualization of the NIPP and NIPP+ approaches prior to implementation. Each intervention arm will receive a 12-week intervention (NIPP or NIPP+) with active monitoring and longitudinal follow ups post intervention at 2, 6, and 12-months post-intervention. The total sample size for the Barrier Analysis will be a maximum of 450 caregivers; for the main intervention, 900 households (300/arm) will be purposely sampled from the randomly selected communities. Respondents for the qualitative portion will be purposely selected.

Analysis: This longitudinal study will collect data from all participants at 3 time points: baseline, endline, and sustainability (12-months post-intervention). The analysis will utilize Intent-to-Treat (ITT) approach using the initial randomization of the treatment arms. Using ITT will allow us to determine the overall impact of having the NIPP vs. NIPP+ vs. control, thus better mimicking real world program implementation and impact. Mixed effects models will be used to determine the role of time-variant and invariant individual (by gender) household, and community characteristics, as well as measures of exposure and integration on key outcome indicators. A difference-in-difference analysis (baseline/endline, baseline/sustainability, endline/sustainability) will also be used to triangulate findings.

Sub-study: a subset of reproductive age women will be purposively selected for enrollment into a validation sub-study that will examine the level of aflatoxin (AFB1-lysine concentration) exposure measured in venous blood compared to capillary blood compared to the innovative SAFE-phone method. This will serve as a validation and calibration sub-study to gauge the accuracy of the SAFE-Phone method compared to venous reference.

ELIGIBILITY:
The inclusion criteria:

* Female circle:

  * Willingness to participate in the group
  * staying in the area for 12 weeks.
  * Have a child under the age of 2 (irrespective of status of malnutrition)
* Male circle inclusion

  * Willingness to participate
  * staying the area for 12 weeks
  * Spouse, brothers and/or other influential male family members of the female caregiver enrolled in the female circle
* Community circle - No specific criteria other than being key community leaders

Exclusion Criteria:

Individuals in households without eligible children (i.e. without a child under age 2), or who will not be present in the selected communities during the intervention and data collection periods and/or who are not willing to participate through the entire 12-week cycle.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1834 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Aflatoxin Exposure in Maize | within 1-month of harvest immediately after the intervention and one year after the intervention.
  aflatoxin in parts per billion in a random sample of maize in a given household's maize supply
Change in E. coli exposure in household | prior to the intervention, immediately after the intervention, and 1 year following the intervention
  e. coli measured in colonies/100 ml

SECONDARY OUTCOMES:
Aflatoxin Exposure in blood serum | immediately after the intervention, and 1 year following the intervention
  venous total (ng/ml) AFB1-lysine adduct concentrations
Aflatoxin Exposure in blood serum | immediately after the intervention, and 1 year following the intervention
  albumin normalized (pg/mg) AFB1-lysine adduct concentrations
Change in Dietary Diversity - mother and child | prior to the intervention, immediately after the intervention, and 1 year following the intervention and 2 and 6-months after the intervention
  24 hours recall applied to standard dietary diversity range

OTHER OUTCOMES:
Change in Mid-upper Arm Circumference | prior to the intervention, immediately after the intervention, and 1 year following the intervention
  cm of mid upper arm circumference taken with standard UNICEF tape
Change in Food Insecurity | prior to the intervention, immediately after the intervention, and 1 year following the intervention
  Household food insecurity and access score (0-27, 72=highly insecure)
Change in weight-for-height z score | prior to the intervention, immediately after the intervention, and 1 year following the intervention
  weight taken with SECA scale and height taken with standard height board applied to WHO growth charts
Maize production | just before exposure to the training and 1 year after training
  acreage planted
Maize production | just before exposure to the training and 1 year after training
  production levels (kg)
Maize production | just before exposure to the training and 1 year after training
  yield (kg/acre)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy P Griswold, MS, Study Director — Tufts University
Locations (1):
- GOAL/Uganda, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
This is undecided, presently
Supporting Information: Study Protocol
Time Frame: The data will be made available via USAID Data Development Library after the first paper has been published.
Access Criteria: Data will be available to the public via the Data Development Library.

REFERENCES:
- [Background] Akombi BJ, Agho KE, Hall JJ, Wali N, Renzaho AMN, Merom D. Stunting, Wasting and Underweight in Sub-Saharan Africa: A Systematic Review. Int J Environ Res Public Health. 2017 Aug 1;14(8):863. doi: 10.3390/ijerph14080863. PMID 28788108
- [Background] Bain R, Bartram J, Elliott M, Matthews R, McMahan L, Tung R, Chuang P, Gundry S. A summary catalogue of microbial drinking water tests for low and medium resource settings. Int J Environ Res Public Health. 2012 May;9(5):1609-25. doi: 10.3390/ijerph9051609. Epub 2012 May 4. PMID 22754460
- [Background] Baoua I.B., Amadou L., Ousmane B., Baributsa D. and Murdock L.L. PICS bags for post-harvest storage of maize grain in West Africa. J. Stored Prod. Res., 58 (2014), pp. 20-28
- [Background] Bauby, AL. and Flachenberg, F. 2014. Achieving sustainability: linking CLTS with other approaches - an example of a thorough WASH intervention in South Eastern Chad. IN: Shaw, R.J., Anh, N.V. and Dang, T.H. (eds). Sustainable water and sanitation services for all in a fast changing world: Proceedings of the 37th WEDC International Conference, Hanoi, Vietnam, 15- 19 September 2014, 5pp
- [Background] Channa H., Ricker-Gilbert J., De Groote H., Marenya P., Bauchet J., Woloshuk C. Assessing Kenyan farmers and traders demand for low cost moisture meters to reduce aflatoxin in maize. Research brief by Purdue University and CIMMYT Kenya.
- [Background] Angood C, Khara T, Dolan C, Berkley JA; WaSt Technical Interest Group. Research Priorities on the Relationship between Wasting and Stunting. PLoS One. 2016 May 9;11(5):e0153221. doi: 10.1371/journal.pone.0153221. eCollection 2016. PMID 27159235
- [Background] Dangour AD, Watson L, Cumming O, Boisson S, Che Y, Velleman Y, Cavill S, Allen E, Uauy R. Interventions to improve water quality and supply, sanitation and hygiene practices, and their effects on the nutritional status of children. Cochrane Database Syst Rev. 2013 Aug 1;2013(8):CD009382. doi: 10.1002/14651858.CD009382.pub2. PMID 23904195
- [Background] Danso J.K., Osekre E.A., Opit G.P., Manu N., Armstrong P., Arthur F.H., Campbell J.F., Mbata G., and McNeill S.G. Post-harvest insect infestation and mycotoxin levels in maize markets in the Middle Belt of Ghana Journal of Stored Products Research 77 (2018) 9-15
- [Background] Davis Jr., Thomas P. Barrier Analysis Facilitator's Guide: A Tool for Improving Behavior Change Communication in Child Survival and Community Development Programs, Washington, D.C.: Food for the Hungry. (2004).
- [Background] ENN. Child wasting and stunting: time to overcome the separation. A Briefing Note for policy makers and programme implementers. Emergency Nutrition Network. June 2018.
- [Background] FTF NIL Africa 2013. Baseline Report. Assessing the linkage between agriculture, food security, nutrition and health among women and children in rural Ugandan households. 66 pages. www.nutritioninnovationlab.org
- [Background] GOAL. 2016. "Implementation guidelines for Nutrition Impact and Positive Practice (NIPP) approach." GOAL, Ireland
- [Background] Hamoudi A, Jeuland M, Lombardo S, Patil S, Pattanayak SK, Rai S. The effect of water quality testing on household behavior: evidence from an experiment in rural India. Am J Trop Med Hyg. 2012 Jul;87(1):18-22. doi: 10.4269/ajtmh.2012.12-0051. PMID 22764286
- [Background] Harding KL, Aguayo VM, Webb P. Factors associated with wasting among children under five years old in South Asia: Implications for action. PLoS One. 2018 Jul 3;13(7):e0198749. doi: 10.1371/journal.pone.0198749. eCollection 2018. PMID 29969457
- [Background] Headey D, Nguyen P, Kim S, Rawat R, Ruel M, Menon P. Is Exposure to Animal Feces Harmful to Child Nutrition and Health Outcomes? A Multicountry Observational Analysis. Am J Trop Med Hyg. 2017 Apr;96(4):961-969. doi: 10.4269/ajtmh.16-0270. Epub 2016 Dec 19. PMID 27994099
- [Background] Khara T, Dolan C. The relationship between wasting and stunting, policy, programming and research implications. Technical Briefing paper. Oxford, UK: Emergency Nutrition Network, 2014. 2.
- [Background] Kikafunda JK, Walker AF, Collett D, Tumwine JK. Risk factors for early childhood malnutrition in Uganda. Pediatrics. 1998 Oct;102(4):E45. doi: 10.1542/peds.102.4.e45. PMID 9755282
- [Background] Korich DG, Mead JR, Madore MS, Sinclair NA, Sterling CR. Effects of ozone, chlorine dioxide, chlorine, and monochloramine on Cryptosporidium parvum oocyst viability. Appl Environ Microbiol. 1990 May;56(5):1423-8. doi: 10.1128/aem.56.5.1423-1428.1990. PMID 2339894
- [Background] Kosinski KC, Kulinkina AV, Abrah AF, Adjei MN, Breen KM, Chaudhry HM, Nevin PE, Warner SH, Tendulkar SA. A mixed-methods approach to understanding water use and water infrastructure in a schistosomiasis-endemic community: case study of Asamama, Ghana. BMC Public Health. 2016 Apr 14;16:322. doi: 10.1186/s12889-016-2976-2. PMID 27076042
- [Background] Lauer JM, Duggan CP, Ausman LM, Griffiths JK, Webb P, Agaba E, Nshakira N, Tran HQ, Gewirtz AT, Ghosh S. Biomarkers of maternal environmental enteric dysfunction are associated with shorter gestation and reduced length in newborn infants in Uganda. Am J Clin Nutr. 2018 Oct 1;108(4):889-896. doi: 10.1093/ajcn/nqy176. PMID 30247538
- [Background] Lauer JM, Duggan CP, Ausman LM, Griffiths JK, Webb P, Bashaasha B, Agaba E, Turyashemererwa FM, Ghosh S. Unsafe Drinking Water Is Associated with Environmental Enteric Dysfunction and Poor Growth Outcomes in Young Children in Rural Southwestern Uganda. Am J Trop Med Hyg. 2018 Dec;99(6):1606-1612. doi: 10.4269/ajtmh.18-0143. PMID 30350765
- [Background] Lauer JM, Duggan CP, Ausman LM, Griffiths JK, Webb P, Wang JS, Xue KS, Agaba E, Nshakira N, Ghosh S. Maternal aflatoxin exposure during pregnancy and adverse birth outcomes in Uganda. Matern Child Nutr. 2019 Apr;15(2):e12701. doi: 10.1111/mcn.12701. Epub 2018 Oct 23. PMID 30242967
- [Background] Luby SP, Rahman M, Arnold BF, Unicomb L, Ashraf S, Winch PJ, Stewart CP, Begum F, Hussain F, Benjamin-Chung J, Leontsini E, Naser AM, Parvez SM, Hubbard AE, Lin A, Nizame FA, Jannat K, Ercumen A, Ram PK, Das KK, Abedin J, Clasen TF, Dewey KG, Fernald LC, Null C, Ahmed T, Colford JM Jr. Effects of water quality, sanitation, handwashing, and nutritional interventions on diarrhoea and child growth in rural Bangladesh: a cluster randomised controlled trial. Lancet Glob Health. 2018 Mar;6(3):e302-e315. doi: 10.1016/S2214-109X(17)30490-4. Epub 2018 Jan 29. PMID 29396217
- [Background] Marshak A, Young H, Bontrager EN, Boyd EM. The Relationship Between Acute Malnutrition, Hygiene Practices, Water and Livestock, and Their Program Implications in Eastern Chad. Food Nutr Bull. 2017 Mar;38(1):115-127. doi: 10.1177/0379572116681682. Epub 2016 Dec 8. PMID 27932595
- [Background] Marshak, A., H. Young, and A. Radday, Water, Livestock, and Malnutrition: Findings from an Impact Assessment of 'Community Resilience to Acute Malnutrition' Programming in the Dar Sila Region of Eastern Chad, 2012-2015. 2016, Feinstein International Center, Tufts University: Medford, MA.
- [Background] Marshak, A., Mazurana, D., Opio, J., Gordon, R., and T. Atim. Tracking change in livelihoods, service delivery, and governance: evidence form a 2013-2015 panel survey in Uganda. ODI Working paper 59. September 2017.
- [Background] Martorell R, Young MF. Patterns of stunting and wasting: potential explanatory factors. Adv Nutr. 2012 Mar 1;3(2):227-33. doi: 10.3945/an.111.001107. PMID 22516733
- [Background] Masset E, Haddad L, Cornelius A, Isaza-Castro J. Effectiveness of agricultural interventions that aim to improve nutritional status of children: systematic review. BMJ. 2012 Jan 17;344:d8222. doi: 10.1136/bmj.d8222. PMID 22251864
- [Background] Murdock L.L., Margam V., Baoua I., Balfe S., and Shade R.E. Death by desiccation: effects of hermetic storage on cowpea bruchids. J. Stored Prod. Res., 49 (2012), pp. 166-170
- [Background] Omotilewa OJ, Ricker-Gilbert J, Ainembabazi JH, Shively GE. Does improved storage technology promote modern input use and food security? Evidence from a randomized trial in Uganda. J Dev Econ. 2018 Nov;135:176-198. doi: 10.1016/j.jdeveco.2018.07.006. PMID 31007346
- [Background] Rogers, Beatrice; Sanchez, Leslie; and Feinstein, Jamie. 2016. Sustaining Development: Results from a Study of Sustainability and Exit Strategies among Development Food Assistance Projects-Honduras Country Study. Washington, DC: FHI 360/Food and Nutrition Technical Assistance III Project (FANTA).
- [Background] Ruel M.T., Quisumbing A.R. and Balagamwalab M. Nutrition-sensitive agriculture: What have we learned so far? Global Food Security 17 (2018) 128-153
- [Background] Schoenbuchner SM, Dolan C, Mwangome M, Hall A, Richard SA, Wells JC, Khara T, Sonko B, Prentice AM, Moore SE. The relationship between wasting and stunting: a retrospective cohort analysis of longitudinal data in Gambian children from 1976 to 2016. Am J Clin Nutr. 2019 Aug 1;110(2):498-507. doi: 10.1093/ajcn/nqy326. PMID 30753251
- [Background] Stobaugh HC, Rogers BL, Rosenberg IH, Webb P, Maleta KM, Manary MJ, Trehan I. Children with Poor Linear Growth Are at Risk for Repeated Relapse to Wasting after Recovery from Moderate Acute Malnutrition. J Nutr. 2018 Jun 1;148(6):974-979. doi: 10.1093/jn/nxy033. PMID 29726948
- [Background] Stobaugh HC, Rogers BL, Webb P, Rosenberg IH, Thakwalakwa C, Maleta KM, Trehan I, Manary MJ. Household-level factors associated with relapse following discharge from treatment for moderate acute malnutrition. Br J Nutr. 2018 May;119(9):1039-1046. doi: 10.1017/S0007114518000363. Epub 2018 Mar 5. PMID 29502542
- [Background] Vella V, Tomkins A, Nviku J, Marshall T. Determinants of nutritional status in south-west Uganda. J Trop Pediatr. 1995 Apr;41(2):89-98. doi: 10.1093/tropej/41.2.89. PMID 7776404
- [Background] Vetter TR, Mascha EJ. Defining the Primary Outcomes and Justifying Secondary Outcomes of a Study: Usually, the Fewer, the Better. Anesth Analg. 2017 Aug;125(2):678-681. doi: 10.1213/ANE.0000000000002224. PMID 28682958
- [Background] Wilson, T. 2007. Perceptions, practices, principles and policies in provision of livestock-water in Africa. Agricultural Water Management, 90 (2007), pp. 1-12
- [Background] Young H., Marshak A. Persistent Global Acute Malnutrition. A discussion paper on the scope of the problem, its drivers and recommendations for policy, practice and research. USA: Feinstein International Center, Tufts University, 2018.
- [Derived] Srinivasan B, Ghosh S, Webb P, Griswold SP, Xue KS, Wang JS, Mehta S. Assessing an aflatoxin exposure biomarker: Exploring the interchangeability and correlation between venous and capillary blood samples. Environ Res. 2022 Dec;215(Pt 2):114396. doi: 10.1016/j.envres.2022.114396. Epub 2022 Sep 23. PMID 36154854
- [Derived] Griswold SP, Marshak A, Fitzpatrick M, Lantagne D, Shoenmakers K, Hebie M, Radday A, De Groote H, Mehta S, Gottlieb G, Webb P, Ghosh S. The One Nutrition in Complex Environments (ONCE) study protocol: a cluster-randomized multi-level multi-sectoral intervention to improve nutrition in Uganda. Trials. 2022 Apr 1;23(1):244. doi: 10.1186/s13063-022-06170-7. PMID 35365180